CLINICAL TRIAL: NCT04479735
Title: Optimizing the Patient Experience: Virtual Reality Goggle Utilization for Venipuncture Distraction - Can we Decrease Anxiety and Pain During This Common Procedure?
Brief Title: Virtual Reality Goggle Utilization for Venipuncture Distraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-11200
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Pain, Procedural
Keywords: virtual reality
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Intervention Model Description: randomized non blinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- VR goggle with venipuncture (Experimental): Virtual reality goggles SamsungGearVR supplied by KindVR will be placed on patients at least 2 min prior to venipuncture. All patients will also receive Lidocaine 2.5%/Prilocaine 2.5% cream at least 60 min prior to venipuncture.
  Interventions: Device: Virtual Reality Goggles
- no VR goggle with venipuncture (No Intervention): Patients will receive Lidocaine 2.5%/Prilocaine 2.5% cream at least 60 min prior to venipuncture but NO virtual reality goggles.

INTERVENTIONS:
Device: Virtual Reality Goggles — Virtual reality goggles will placed at least 2 min prior to venipuncture to deteremine if it mitigates perceived anxiety or perceived pain scores.
  Arms: VR goggle with venipuncture

SUMMARY:
This is a randomized non-blinded trial evaluating the effect of virtual reality goggles on perceived pain and anxiety scores during venipuncture on hospitalized children ages 5-21. We will randomized patients to either standard of care (including Lidocaine 2.5%/Prilocaine 2.5% cream as a topical anesthetic 60-240 minutes prior to venipuncture) or standard of care plus virtual reality goggles.

DETAILED DESCRIPTION:
Study personnel will identify patients on CHAM 6 and CHAM 8 scheduled for lab draw prior to child life rounds and subsequently ask the health care providers if there are any patients that are not developmentally or physically appropriate to use the VR equipment. They will then screen and consent the patients approximately 1 hour prior to the Child Life rounds (see appendix A & B). Patients aged 12-17 years old who are able to read the form will be asked to fill out an assent form (see appendix C) and patients aged 5-12 years old and those unable to read the form will be read the assent form to ensure verbal assent. Those patients who consent to the study will be randomized to a VR arm and non VR arm using computer generated randomization. Lidocaine 2.5%/Prilocaine 2.5% cream will be placed on all patients that have consented to the study by the patient's nurse if they don't already have it applied. After consent and assurance of topical anesthetic application, a brief demographic questionnaire (see appendix D) will also be completed. For efficiency and feasibility, two study personnel will screen and consent families, assist with VR set up and removal, and conduct post procedure assessment.

ELIGIBILITY:
Inclusion Criteria:

patients aged 5-21 years old admitted to the 6th floor of the inpatient unit who are scheduled for a venipuncture during morning phlebotomy rounds

Exclusion Criteria:

Patients developmentally or physically not appropriate to use the VR equipment as determined by their parent, guardian or healthcare provider, if there is discomfort related to wearing the goggles (for example: recent neurosurgery, migraines, hardware on head), patient have photosensitive seizures or infectious concern such as scabies, lice, COVID-19 that can't reliably be disinfected.

Patient (>18) or Parent or guardian (for patient < 18) that does not speak English, Spanish or Arabic will be excluded.

If patient refuses Lidocaine 2.5%/Prilocaine 2.5% cream use they will also be excluded from the study.

-

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived Pain Scale | Approximately 1 hour prior to venipuncture and again immediately after venipuncture
  Change in perceived pain from pre-venipuncture to post-venipuncture (during the blood draw) will be assessed using the Wong-Baker FACES Pain Rating scale. Children, or parents on behalf of children, will be asked to communicate the severity of the pain the child is experiencing using the FACES scale which contains a series of 6 different facial expressions correlated to numbers (i.e., 0, 2, 4, 6, 8, 10) ranging from a happy face at "0" indicating "no hurt" to a crying face at "10" indicating "hurts worst." Higher scale scores signify worse pain severity. Change in group mean FACES scale scores will be summarized by study arm and subsequently analyzed using Wilcoxon signed rank test for paired data.

SECONDARY OUTCOMES:
Change in Anxiety Scores | Approximately 1 hour prior to venipuncture and again immediately after venipuncture
  Change in anxiety from pre-venipuncture to post-venipuncture (during the blood draw) will be assessed using the Visual Analog Scale (VAS). Children, or parents on behalf of children, will be asked to estimate the level of anxiety the child is having by marking their estimate on a visual 0-to-100 millimeter (mm) line ranging from "0" (=Not at all Anxious) to "100" (=Extremely Anxious). The line increases by increments of "1" from left to right. A score of ≥ 30mm is considered anxious. Change in anxiety scores will be summarized by study arm using basic descriptive statistics and subsequently analyzed using Wilcoxon signed rank test for paired data.
Change in Heart Rate | Approximately 1 hour prior to venipuncture and again immediate after venipuncture
  Change in HR from pre-venipuncture to post-venipuncture will be evaluated for those patients on a cardiac monitor. Increased heart rate can be associated with increases in pain and anxiety. Group mean changes in heart will be summarized by study arm and subsequently analyzed using Wilcoxon signed rank test for paired data.
Change in Level of simulator sickness | Approximately 1 hour prior to venipuncture and again immediately after venipuncture
  Change in Level of simulator sickness from pre-venipuncture (pre-placement of Virtual Reality goggles) to post-venipuncture (removal of VR goggles) will be assessed using a Simulator Sickness Questionnaire. The survey consists for 4 questions related to the possible side effects of using the VR goggles. Children, or parents on behalf of children, will be asked to respond to the following 4 questions on a scale ranging from 1-10: Does your head hurt? Do your eyes hurt? Do you have an upset stomach? Do you feel dizzy? Total scores will be summed for an overall possible scoring range of 4-40 with higher scores indicating worse sickness symptoms. Change in simulator sickness scores will be summarized by study arm.
Pre-venipuncture anxiety scores in participants with prior hospitalizations or prior medical problems. | Baseline
  Level of pre venipuncture anxiety scores in participants with prior hospitalizations or prior medical problems will be evaluated. Anxiety scores will be collected using the VAS tool. Children, or parents on behalf of children, will be asked to estimate the level of anxiety the child is having by marking their estimate on a visual 0-to-100mm line ranging from "0" (=Not at all Anxious) to "100" (=Extremely Anxious). The line increases by increments of "1" from left to right. A score of ≥ 30mm is considered anxious. Prior hospitalization data and prior medical problem information will be extracted via chart review. Anxiety scores will be summarized by study arm using basic descriptive statistics. An independent t test will be used to asses whether anxiety scores are normally distributed or Mann U test if not normally distributed.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney A McNamara, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No